CLINICAL TRIAL: NCT00342836
Title: Immunohistochemical Analysis of Human Transbronchial Biopsy Specimens Collected in a Phase I Chemoprevention Trial of Myo-Inositol in Heavy Smokers Conducted Outside the Intramural NCI Program
Brief Title: Analysis of Tissues From Patients in Trial of Myo-Inositol to Prevent Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999905146; 05-C-N146; NCT00899730 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2007-03-23 (Estimated); Status verified 2006-02

CONDITIONS: AKT
Keywords: Akt; Immunohistochemistry; Myoinositol; Bronchial Specimens; Phosphorylation

INTERVENTIONS:
Procedure: Akt levels

SUMMARY:
This study will examine tissue specimens from patients participating in a trial of high-dose myo-inositol to prevent lung cancer. The trial, conducted at the British Columbia Cancer Agency-Vancouver Cancer Center (BCCA-VCC), includes people who have pre-cancerous changes in the air passages of their lungs.

The BCCA-VCC trial was designed to determine side effects of taking large amounts of the food supplement myo-inositol for longer than a month and if the supplement can help smokers stop smoking.

The current study will look at the levels of a substance called Akt in tissue samples obtained from air passages of subjects in the BCCA-VCC trial. Akt is activated by tobacco components and can be found in lung tumor specimens and pre-cancerous lesions. Myo-inositol may affect Akt levels and help prevent progression of pre-cancerous lesions to cancer.

People participating in the BCCA-VCC phase 1 myo-inositol trial are eligible for this study. Tissue samples obtained from air passages of these patients during their participation in that study will be sent to the National Cancer Institute for analysis of Akt levels.

DETAILED DESCRIPTION:
Human transbronchial biopsy specimens collected under protocol study numbers CDR0000302633; BCCA-U98-0411; BCCA-C02-0298 will be immunohistochemically stained for activated Akt using phospho-specific antibodies. These samples are part of a phase I chemoprevention trial of myo-inositol being conducted in Vancouver, BC by the British Columbia Cancer Agency in collaboration with the National Cancer Institute (NCI). The transbronchial specimens will be sent to the NCI for analysis of activated AKT. The study aims to determine whether myo-inositol, a putative inhibitor of the upstream kinase phosphatidylinositol 3-kinase, can alter activated Akt levels in smokers with bronchial dysplasia.

ELIGIBILITY:
* INCLUSION CRITERIA:

Any patients entered into phase 1 myo-inositol trial are eligible for inclusion, provided that they have consented to tissue analysis in the original consent form.

EXCLUSION CRITERIA:

None anticipated at this time.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-04

CONTACTS AND LOCATIONS:
Locations (1):
- British Columbia Cancer Agency (BCCA), Vancouver, Canada

REFERENCES:
- [Background] Hecht SS, Kenney PM, Wang M, Upadhyaya P. Dose-response study of myo-inositol as an inhibitor of lung tumorigenesis induced in A/J mice by benzo. Cancer Lett. 2001 Jun 10;167(1):1-6. doi: 10.1016/s0304-3835(01)00454-2. PMID 11323092